CLINICAL TRIAL: NCT04280471
Title: An Open-Label Phase 1 Pilot Study: Fecal Microbiota Transplantation (FMT) in Severe Acute Gut Graft-Versus-Host Disease Patients
Brief Title: Fecal Microbiota Transplantation for the Treatment of Severe Acute Gut Graft-Versus-Host Disease
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was not opened
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-001736; NCI-2020-00211 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19-001736 (Other: UCLA / Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2020-02-05; First posted 2020-02-21 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2022-11

CONDITIONS: Acute Graft Versus Host Disease; Gastrointestinal Tract Acute Graft Versus Host Disease; Severe Gastrointestinal Tract Acute Graft Versus Host Disease; Steroid Resistant Gastrointestinal Tract Acute Graft Versus Host Disease
Keywords: Gut GvHD; FMT
MeSH Terms: interventions — Fecal Microbiota Transplantation; Parturition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (OpenBiome FMT capsule DE) (Experimental): Patients ingest OpenBiome FMT Capsule Dose Extended (DE) orally for two consecutive days. One dose is equivalent to the ingestion of 30 capsules and thus each day the patient will ingest 15 capsules. If no response is noted after 7 days, patients may receive a second dose of FMT for an additional 2 days.
  Interventions: Drug: Fecal Microbiota Transplantation Capsule

INTERVENTIONS:
Drug: Fecal Microbiota Transplantation Capsule — Receive OpenBiome FMT Capsule DE PO
  Other Names: Fecal Microbiota Preparation Delivery Capsule; FMPCapDE; FMT Capsule DE; FMT Capsule Delivery; FMT DE Capsule

SUMMARY:
This phase I trial studies the side effects of using an investigational procedure (fecal microbiota transplantation [FMT]) in treating patients with severe acute gut graft-versus-host-disease. The purpose of a fecal microbiota transplantation is to use feces from a healthy human donor to replace the abnormal gut bacteria in the recipient. One of the side effects of a stem cell transplant is the development of graft-versus-host disease (GvHD) in several organs including gut. GvHD is caused by the donated bone marrow or peripheral blood cells recognizing the recipient's body as foreign and attacking it. Acute gut GvHD is one of the leading causes of death after transplant. Recently, studies have shown that patients with reduced intestinal bacterial diversity in their stool during acute gut GvHD have higher overall mortality rates. The information learned from this study may offer FMT as a promising therapy for the treatment of severe acute gut graft-versus-host-disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. For safety evaluation, episodes of microbial bloodstream infection attributed to fecal microbiota transplantation (FMT) within the first 7 days after start of each FMT administration.

II. For tolerability evaluation, subject must ingest 50% of one dose of FMT product without grade 3 or higher adverse events (AEs) within the first 7 days post-FMT.

SECONDARY OBJECTIVE:

I. To collect stool, oral swabs and blood specimens for future studies to define bacterial taxa diversity, microbial translocation as well as metabolomic and proteomic changes associated with the development of graft versus host disease (GvHD).

II. For clinical efficacy, > 50% of subjects with at least 1 stage of gut GvHD improvement by 8 weeks after the first dose of FMT.

OUTLINE:

Patients ingest OpenBiome FMT Capsule Dose Extended (DE) orally for two consecutive days. One dose is equivalent to the ingestion of 30 capsules and thus each day the patient will ingest 15 capsules. If no response is noted after 7 days, patients may receive a second dose of FMT for an additional 2 days. Standard treatment for gut GvHD will continue during this time.

After completion of study treatment, patients are followed for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who received an allogenic hematopoietic stem cell transplantation (HSCT)
* Acute GvHD defined as experiencing GvHD symptoms starting prior to day +100 after HSCT
* Gut GvHD defined as subjects experiencing GvHD symptoms consistent with stage 3 or stage 4 by Center for International Blood and Marrow Transplant Research (CIBMTR) staging:

  * Stage 3 acute gut GvHD subjects having 1500-1999 mL stool per day
  * Stage 4 subjects having greater than 2 liters of stool per day and/or severe abdominal cramping, bleeding or ileus
* Steroid-refractory acute gut GVHD defined as progression of symptoms after 3 days of systemic steroids (> 1 mg/kg/day methylprednisolone) or steroid-resistant acute gut GvHD defined stable symptoms after 5 days of systemic steroids (> 1 mg/kg/day methylprednisolone)
* Able to swallow capsules without aspiration or dysphagia
* Ability to understand the written informed consent and the willingness to sign the consent and accept the risk of receiving unrelated donor stool

Exclusion Criteria:

* Absolute neutrophil count < 500 cells/uL
* Presence of recurrent Clostridium difficile infection
* Presence of ileus or toxic megacolon
* History of multi-drug resistant stool pathogen
* History of inflammatory bowel disease (i.e Crohn's disease or ulcerative colitis)
* Uncontrolled and active systemic infection from bacteria, virus or fungus
* Human immunodeficiency virus (HIV)-positive subjects
* Quantifiable cytomegalovirus (CMV) and/or Epstein-Barr virus (EBV) evaluated by polymerase chain reaction (PCR) after hematopoietic stem cell transplantation (HSCT) and after neutrophil engraftment defined as absolute neutrophil count (ANC) > 500 cells/uL
* Hemodynamically unstable
* Active gastrointestinal bleed
* Pregnant and/or breastfeeding women
* Dysphagia due to oropharyngeal, esophageal, functional, neuromuscular (e.g. stroke, multiple sclerosis, amyotrophic lateral sclerosis [ALS]) or subject shows evidence of dysphagia when the 'safety test' capsule is administered
* Delayed gastric emptying syndrome
* Known chronic aspiration
* Subjects with a history of significant allergy to foods
* Subjects with allergies to sodium chloride, glycerol, theobroma oil, hide bovine gelatin, sodium lauryl sulfate, colorants Federal Food, Drug, and Cosmetic Act (FD&C), or titanium dioxide, all ingredients generally recognized as safe (GRAS)
* History of previous gastrointestinal surgery
* Subjects who are receiving other investigational agents for treatment of gut GvHD

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 6 months
  For safety evaluation, episodes of microbial bloodstream infection attributed to fecal microbiota transplantation (FMT) within the first 7 days after start of each FMT administration. For tolerability evaluation, at least 60% of subjects able to ingest 50% of one dose of FMT without grade 3 or higher adverse events (AEs) within the first 7 days post-FMT. Subjects will be monitored via assessment of gut graft versus host disease (GvHD) staging and adverse events will be performed bi-weekly for the first 4 weeks after the first dose of FMT, weekly during the hospitalization and monthly up to six months after hospital discharge.

SECONDARY OUTCOMES:
Collection of stool, oral swabs and blood specimens to define bacterial taxa diversity, microbial translocation as well as metabolomic and proteomic changes associated with the development of graft versus host disease (GvHD) | Up to 6 months
  Alpha diversity metrics will be compared between time points mixed effect regression models. Multivariate differences will be calculated using permutational multivariate analysis of variance (PERMANOVA). Differential abundance techniques will be used to compare taxa over time using DESeq2 package. DESeq2 models taxa counts with a negative binomial model. To look specifically at before and after FMT, we will apply multivariate techniques such as principal coordinate analysis (PCoA) to identify parameters that are affected positively by FMT and to determine whether these differences persist over time. The PERMNOVA technique will be applied to survey population-level differences before & after FMT. We will use the Benjamini-Hochberg false discovery rate (FDR) to account for multiple hypothesis testing.
GvHD improvement | Up to 8 weeks after the first dose of FMT
  Clinical efficacy will be defined as > 50% of subjects with at least 1 stage of gut GvHD improvement by 8 weeks after the first dose of FMT.

CONTACTS AND LOCATIONS:
Overall Officials: Grace Aldrovandi, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States